CLINICAL TRIAL: NCT04959617
Title: Multi-center Application Study of Quantitative FIT Technology for Colorectal Cancer Screening in Chinese Physical Examination Population
Brief Title: Multi-center Application of Quantitative FIT Technology in Colorectal Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); The Second Hospital of Anhui Medical University (Other); The First Hospital of Jilin University (Other); Sino-Japanese Friendship Hospital of Jilin University (Unknown); First Hospital of China Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The Second Hospital of Hebei Medical University (Other); The First Hospital of Hebei Medical University (Other); Jiangsu Provincial People's Hospital (Other); The Second Hospital of Nanjing Medical University (Other); Jiangxi Provincial People's Hopital (Other); Second Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Harbin Medical University (Other); Peking Union Medical College Hospital (Other); Shenzhen People's Hospital (Other); Guangdong Provincial People's Hospital (Other); Tongji Hospital (Other); First Affiliated Hospital of Suzhou Medical College (Other); Chinese PLA General Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital of Inner Mongolia Medical College (Unknown); Bethune International Peace Hospital (Other); Xinqiao Hospital of Chongqing (Other); Renmin Hospital of Wuhan University (Other); The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-181
Record Dates: First submitted 2021-07-11; First posted 2021-07-13 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer Screening Fecal Immunochemical Test

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Quantitative Fecal Immunochemical Test (qFIT) — The study only included quantitative FIT examination in the general physical examination population over 30 years old.

SUMMARY:
In order to control the incidence of colorectal cancer, improve the level of early diagnosis and early warning the occurrence of colorectal cancer, it is very necessary for us to explore the threshold value of FIT positive judgment in line with the Chinese population, and further contribute to the establishment of a colorectal cancer screening pathway suitable for Chinese healthy population

DETAILED DESCRIPTION:
Feces were collected for quantitative FIT test. Those with positive results were further examined by colonoscopy. By comparing with pathological results of colonoscopy, the sensitivity, specificity, positive predictive value and negative predictive value of quantitative FIT technology for the diagnosis of colorectal tumors were confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people aged 30 years and planning to undergo colonoscopy;
2. No history of gastrointestinal tumor;
3. No ulcerative colitis or Crohn's disease;
4. No gastrointestinal hemorrhagic disease;
5. No history of gastrointestinal surgery, able to understand and willing to sign informed consent.

Exclusion Criteria:

1. Other serious diseases of the digestive tract, such as Crohn's disease ulcerative colitis;
2. Patients with gastric and esophageal cancer and other malignant tumors;
3. Unable to cooperate after communication;
4. Subjects who have received radiotherapy and chemotherapy;
5. Other researchers believe that they are not suitable for inclusion in this clinical trial, such as mental illness patients, critical patients, pregnant women, illiterate minors, cognitive impairment PI, students of the researcher, PI, affiliated research units of the co-investigator or employees of the sponsor, etc

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy physical examination person over 30 years of age
Sampling Method: Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2019-01-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of quantitative FIT | 1year
  The sensitivity of quantitative FIT application in Chinese physical examination population
Specificity of quantitative FIT | 1year
  The specificity of quantitative FIT application in Chinese physical examination population

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided